CLINICAL TRIAL: NCT00678496
Title: Computerised Cognitive Behavioural Therapy for Treatment of Depression in MS (CoSMoS): Clinical Trial Pilot Study
Brief Title: Cognitive Behavioural Therapy Software for the Treatment of Depression in People With Multiple Sclerosis
Acronym: CoSMoS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other); Walton Centre NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112276; EudraCT number: 2008-001039-37; MS Society: 845/06
Record Dates: First submitted 2008-05-14; First posted 2008-05-15 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-09

CONDITIONS: Depression; Multiple Sclerosis
Keywords: CBT-software; Computerised Cognitive Behavioural Therapy; CCBT; Cognitive Therapy; Therapy, Computer-Assisted; Depression; Multiple Sclerosis
MeSH Terms: conditions — Depression; Multiple Sclerosis | interventions — Therapeutics; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CBT software delivered at home or in a primary care facility (n=12)
  Interventions: Other: CBT Software
- 2 (Other): Treatment as usual (n=12)
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: CBT Software — Beating the Blues is a CBT-based software package for patients with anxiety and/or depression. The CBT strategies used include: identifying thinking errors, challenging automatic negative thoughts, modifying attributional style and identifying core beliefs. The behavioural techniques used include graded exposure, sleep management, problem solving, task breakdown and activity scheduling. The programme consists of a 15 minute "Introduction to Therapy" video plus eight computer-interactive sessions of approximately 50 minutes each in duration. Each session consists of a mix of cognitive and behavioural strategies, which are customised to the patient's individual problems. The eight computer sessions are designed to be taken weekly, or thereabouts, and each session builds on the previous one.
  Other Names: Ultrasis Beating the Blues; Beating the Blues
  Arms: 1
Other: Treatment as usual — Participants in the usual care arm are asked to refrain from accessing psychological services during their participation in the study, but may be prescribed anti-depressants or referred to a counsellor by their general practitioner.
  Other Names: Waiting list; Usual care; Treatment As Usual (TAU)
  Arms: 2

SUMMARY:
Guidance issued by the United Kingdom (UK) National Institute for Health and Clinical Excellence (NICE) recommends the use of computerised cognitive behavioural therapy (CCBT) 'Beating the Blues' (BtB) in treatment of depression. However CCBT has not been designed specifically for use by people with Multiple Sclerosis (MS) and may not be effective or appropriate for use by people with physical disabilities or cognitive symptoms. There would therefore be value in conducting a trial of the effectiveness of CCBT for depression in people with MS. The aim of this pilot study is to test the feasibility of a randomised control trial (RCT) of CCBT for depression in people with MS. The objective is to undertake a pilot RCT of comparison of CCBT with usual care including 3 month follow up to identify a realistic patient recruitment rate and provide reliable estimates of other parameters needed for designing a definitive RCT including the sample size. Other outcomes to be measured include estimates of the effect on depression and quality of life. Participants will be assessed as experiencing clinical levels of depression and be recruited from two participating MS Centres. The outcomes of the study will be (1) preliminary indication of the impact of CCBT on depression in MS; and, (2) a well researched protocol for a definitive RCT of the effectiveness of CCBT in treating depression in people with MS.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+
* Diagnosis of MS confirmed by neurologist
* Beck Depression Inventory-II score of at least 14 on two consecutive occasions
* Not currently or within past three months receiving any treatment from a psychologist, psychotherapist or psychiatrist.
* Willingness to be randomised to CCBT, at home or primary care facility or treatment as usual.

Exclusion Criteria:

* Unable to read or write English
* Beck Depression Inventory score of at least 29 on two consecutive occasions
* Active suicidal ideas
* Current or life-time diagnosis of any of the following:

  * psychosis
  * organic mental disorder;
  * alcohol or drug dependency
* Kurtzke Expanded Disability Status Scale (EDSS) score of 8.5 or above
* Unable to use the CCBT package due to physical disability
* Unable to use the CCBT package due to cognitive symptoms (mini-mental state of 20 below or if, in the opinion of the study psychologist, the individual would be unlikely to benefit from CCBT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2010-01-31 (Actual); Study Completion 2010-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L Cooper, PhD, Principal Investigator — University of Sheffield; Glenys D Parry, PhD, Study Chair — University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We reached our recruitment target on 30 July 2009 (in 281 days; 2.6 participants/month) after adding a second centre (The Walton Centre National Health Service (NHS) Foundation Trust, Liverpool).
Pre-assignment Details: Participants were invited to take part via clinic mailouts. Responders were excluded if their Beck Depression Inventory score was too high, too low, if they were under the care of a psychiatrist, or were not resident within the boundaries of participating primary care trusts (UK NHS commissioning bodies 2001-2013), or if they refused consent.
Groups:
- Computerised CBT Using 'Beating the Blues'® (Ultrasis Ltd): CBT software (n=12). Beating the Blues® consists of eight computer-interactive sessions, of approximately 50 minutes each in duration, designed to be taken weekly.
- Treatment as Usual: Treatment as usual (n=12). The research protocol did not manualise or restrict treatment as usual, but a client service receipt inventory was used at baseline, 8 weeks and 21 weeks to identify concomitant medication and service use in both arms.
Period: Overall Study
Arm/Group | Computerised CBT Using 'Beating the Blues'® (Ultrasis Ltd) | Treatment as Usual
Started | 12 | 12
Completed 8 Weeks Follow-up | 9 | 12
Completed | 10 | 8
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- CBT Software: CBT using 'Beating the Blues'® software (Ultrasis Ltd). Beating the Blues® consists of eight computer-interactive sessions, of approximately 50 minutes each in duration, designed to be taken weekly. Each session consists of a mix of cognitive and behavioural strategies, which the user customises to their individual problems.
- Treatment as Usual: Treatment as usual. The research protocol did not manualise or restrict treatment as usual, but a client service receipt inventory was used at baseline, 8 weeks and 21 weeks to identify concomitant medication and service use in both arms.
- Total: Total of all reporting groups
Arm/Group | CBT Software | Treatment as Usual | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (7.7) | 42 (7.0) | 45 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 1 | 5 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Expanded Disability Status Scale (EDSS) score [Mean (Standard Deviation); unit: units on a scale] — Kurtzke Expanded Disability Status Scale (EDSS) tool for quantifying MS-related disability. Scale of 0-10, with 10 being the highest disability. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability.
  units on a scale | 4.8 (1.7) | 3.6 (1.8) | 4.2 (1.8)
BDI total score (0 weeks) [Mean (Standard Deviation); unit: units on a scale] — Beck Depression Inventory II-21 Item (BDI-II) - a self-report measure of severity of symptoms of depression. This is scored by summing the ratings for the 21 items. Each item is rated on a 4-point scale ranging from 0 to 3. The maximum total score is 63 (severe depression).
  units on a scale | 21 (4.0) | 23 (5.2) | 22 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-reported Symptoms of Depression, as Measured by Total BDI-II Score
Description: Beck Depression Inventory II-21 Item (BDI-II) - a self-report measure of severity of symptoms of depression. This is scored by summing the ratings for the 21 items. Each item is rated on a 4-point scale ranging from 0 to 3. The maximum total score is 63 (severe depression).
  The study reports change from baseline at 21 weeks.
Time Frame: 21 weeks
Population: There may be different numbers of patients analysed at 8 weeks and 21 weeks, as patients may have dropped out, or there may have been missing information at 8 weeks meaning that the score could not be calculated, but the patient was still followed up at 21 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CCBT: Ultrasis - Beating the Blues® is a computer-interactive programme for the treatment of anxiety and depression. It is based on cognitive behavioural therapy (CBT), which helps patients to identify and change unhelpful ways of thinking and to learn more effective ways of solving problems.
- Treatment as Usual: The research protocol did not manualise or restrict treatment as usual. A client service receipt inventory was used at baseline, 8 weeks and 21 weeks to identify concomitant medication and service use in both arms.
Arm/Group | CCBT | Treatment as Usual
Number analyzed (Participants) | 10 | 12
units on a scale
  8 weeks: number analyzed (Participants) | 9 | 12
  8 weeks | -5.33 (4.7) | -1.17 (8.1)
  21 weeks | -2.00 (5.1) | 0.25 (8.8)

2. Secondary Outcome: Change in Disease-specific Quality of Life, Measured on the Multiple Sclerosis Impact Scale-29 Item (MSIS-29)
Description: The Multiple Sclerosis Impact Scale (MSIS-29) is a 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of MS on day-to-day life in the past two weeks. All items have 5 response options: 1 "not at all" to 5"extremely". Each of the two scales are scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates greater impact of disease on daily function (worse health).
  This study measured the change from baseline at 8 weeks and 21 weeks.
Time Frame: Eight weeks or on completion of CCBT (whichever is later), and three months thereafter.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CCBT: CCBT using 'Beating the Blues'® (Ultrasis Ltd). Beating the Blues® consists of eight computer-interactive sessions, of approximately 50 minutes each in duration, designed to be taken weekly. Each session consists of a mix of cognitive and behavioural strategies, which the user customises to their individual problems.
Arm/Group | CCBT | Treatment as Usual
Number analyzed (Participants) | 9 | 11
units on a scale
  Psychological - 8 weeks: number analyzed (Participants) | 8 | 11
  Psychological - 8 weeks | -5.88 (9.5) | 0.18 (5.1)
  Psychological - 21 weeks: number analyzed (Participants) | 9 | 10
  Psychological - 21 weeks | -4.33 (8.0) | -2.60 (5.6)
  Physical - 8 weeks: number analyzed (Participants) | 8 | 11
  Physical - 8 weeks | -7.00 (12.9) | -1.82 (7.8)
  Physical - 21 weeks: number analyzed (Participants) | 9 | 10
  Physical - 21 weeks | -7.89 (12.3) | -2.20 (11.0)

ADVERSE EVENTS:
Groups:
- CCBT Using 'Beating the Blues'® (Ultrasis Ltd): CBT software (n=12). Beating the Blues® consists of eight computer-interactive sessions, of approximately 50 minutes each in duration, designed to be taken weekly.
Arm/Group | CCBT Using 'Beating the Blues'® (Ultrasis Ltd) | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CCBT Using 'Beating the Blues'® (Ultrasis Ltd) (N=8) | Treatment as Usual (N=10)
Broken arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Deemed not related with the intervention, not related to natural history of MS and recovered with no sequelae.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No